CLINICAL TRIAL: NCT05385705
Title: A Phase Ib Study With a Safety lead-in Cohort and Expansion Phase, of the Safety, Tolerability, Biological Effect, and Efficacy of Allogenic Natural Killer Cells in Combination With Trastuzumab and Pertuzumab in Adult Patients With Refractory Metastatic Her2 Positive Breast Cancer
Brief Title: A Study of Allogenic Natural Killer Cells in Combination With Trastuzumab and Pertuzumab in Adult Patients With Refractory Metastatic Her2 Positive Breast Cancer. NK-ACT-BC_2020
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other); Puerta de Hierro University Hospital (Other); Hospital del Mar (Other); Banc de Sang i Teixits (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHIO20002
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Trastuzumab; pertuzumab; Interleukin-2

STUDY DESIGN:
Intervention Model Description: This is an open label, multi-center, proof of concept, phase Ib trial.
  A total of 6 patients will be included in the safety lead-in phase. If signs of both clinical and biological activity are seen, and no more than 1 TLT is observed in those first 6 patients, the study will expand with 14 additional patients (expansion phase).
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: NKs (Experimental): Subjects will be treated with cyclophosphamide single dose between days -5 and -3 before the NK-cell infusion. On Day 1 single loading doses of trastuzumab (8mg/kg iv) and pertuzumab (840 mg iv) will be administered followed by maintenance doses of 6mg/kg and 420mg respectively, every three weeks. After that, NK infusion will be done on day 2 and that will be followed by administration of IL-2 on day 2, 4 and 6 as a subcutaneous dose of 5x105 UI/m2.
  Interventions: Drug: Cyclophosphamide; Drug: Trastuzumab; Drug: Pertuzumab; Biological: NK cells; Drug: Interleukin-2

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide at a single dose of 600mg/m2 IV between days -5 and -3 before NK cell infusion for preconditioning the tumoral microenvironment by reducing the levels of lymphocyte T regulators (Tregs FOXP3+, CD3+, CD4+, CD25+).
Drug: Trastuzumab — Trastuzumab at a dose of 8mg/kg IV for the loading dose on Day 1, and 6mg/kg IV for the maintenance dose every 3 weeks (Q3W).
Drug: Pertuzumab — Pertuzumab at a dose of 840mg IV for the loading dose on Day 1, and 420 mg IV for the maintenance dose every 3 weeks (Q3W).
Biological: NK cells — NK product is a cellular investigational product comprising a live cell suspension of allogenic NK cells derived from a compatible donor that will be infused on Day 2.
Drug: Interleukin-2 — IL-2 (Proleukin) will be administered on Day 2 (within 24h after NK infusion), 4 and 6 as a subcutaneous dose of 5x105 UI/m2, following the label instructions.

SUMMARY:
Breast cancer is the second most common invasive malignancy and the leading cause of cancer-related mortality in women. Overexpression of human epidermal growth factor receptor 2 (HER2) is observed in approximately 20% of breast cancers.

Trastuzumab provided patients with HER2 overexpressing breast cancer a better outcome than chemotherapy alone. Trastuzumab and pertuzumab exert part of their activity based on antibody-dependent cell-mediated cytotoxicity (ADCC), mediated by natural killer (NK) cells.

Trastuzumab (Herceptin®) is a recombinant DNA-derived humanized monoclonal antibody that selectively binds with high affinity to the extracellular domain of the human epidermal growth factor receptor 2 (HER2). Inhibits the proliferation of human tumor cells that overexpress HER2 and to mediate antibody-dependent cellular cytotoxicity (ADCC).

Pertuzumab (Perjeta®) is a fully humanized monoclonal antibody and, like trastuzumab, is directed against the extracellular domain of HER2. It differs from trastuzumab because they bind to different domains. Due to their distinct mechanisms of action, the combination of pertuzumab and trastuzumab, is hypothesized to have complementary roles in treating HER2-overexpressing diseases.

Natural killer cells are lymphocytes arising from CD34+ hematopoietic progenitor cells in the bone marrow. NK cells are identified as CD3-, CD56+ lymphocytes. These cells were identified on the basis of their ability to lyse tumor cells without prior sensitization. NK function is also regulated by cytokines such as IL-2, IL-15, IL-12 and IL-18.

Our hypothesis is that the effect of trastuzumab and pertuzumab can be improved by regulating the efficiency of the ADCC activity through the infusion of ex-vivo activated allogenic NK cells.

Objetives:

Primary: To assess the safety and the tolerability of NK-ACT and trastuzumab/pertuzumab when used in combination.

Secondary: To evaluate the initial clinical activity of NK-ACT concomitant with trastuzumab/pertuzumab.

Exploratory Objectives: In vivo human NK cell biology:

* To describe the mechanisms of action of the combination of ICTP and rastuzumab/pertuzumab.
* To assess the biomarkers that might act as indicators of the immunemodulatory effect and anti-tumor activity of the combination.

DETAILED DESCRIPTION:
This is an open label, multi-center, proof of concept, phase Ib trial.

A total of 6 patients will be included in the safety lead-in phase. If signs of both clinical and biological activity are seen, and no more than 1 TLT is observed in those first 6 patients, the study will expand with 14 additional patients (expansion phase).

Enrollment - 24 months

Duration - 35 months

During the lead-in phase and the expansion phase, a staggered enrollment will be employed. In the lead-in phase, the subsequent patient will start the treatment after the TLT period completion (28 days) of the previously treated patient.

In the expansion cohort, the patients will be dosed successively with a safety monitoring interval of at least 48 hours between the last subcutaneous administration of IL-2 in the previous patient and the first administration of intravenous cyclophosphamide (D-5) in the subsequent patient.

Study treatment:

Cyclophosphamide at a single dose of 600mg/m2 IV between days -5 and -3 before NK cell infusion.

Trastuzumab at a dose of 8mg/kg IV for the loading dose, and 6mg/kg IV for the maintenance dose every 3 weeks (Q3W).

Pertuzumab at a dose of 840mg IV for the loading dose, and 420 mg IV for the maintenance dose every 3 weeks (Q3W)

NKs at a minimum dose of 5x107 NKc and at a maximum dose limit of 5x108 NKc.

IL-2 at a dose of 5x105 UI/m2, on day 2, 4, and 6 after NK infusion.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Histologically confirmed locally advanced and/or metastatic breast adenocarcinomas that have progressed on standard therapy (must have received pertuzumab, trastuzumab, and ado-trastuzumab emtansine in the neoadjuvant, adjuvant, or metastatic setting) and have received at least two lines of therapy in the metastatic setting. Prior neoadjuvant or adjuvant therapy presenting relapse within 6 months of completion will be considered as a line of treatment for metastatic disease. Hormonal therapies will not be considered as previous lines of therapy. Eligible patients must have progressed while on or following the most recent line of therapy.
2. Patient's provision of signed Informed Consent.
3. Patient has potential allogenic donors (alive parents, siblings, patient´s couple or children aged ≥ 18 years) who provide signed Donor Informed Consent. A trial physician will address the suitability of the identified allogenic relative as an optimal candidate.
4. Age ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Life expectancy ≥ 3 months.
7. Ability to comply with the protocol requirements.
8. Patients must have clinically and/or radiographically documented measurable disease. At least one lesion must be measurable as per RECIST v.1.1. Previously irradiated lesions must not be counted as target lesions unless there has been demonstrated progression in the lesion and no other target lesions are available.

   Tumors must be accessible for pre-planned biopsies. Lesions that are intended to be biopsied must not be counted as target lesions.
9. Adequate hematologic and organ function defined by the following laboratory results obtained within 7 days prior to the first study treatment (cyclophosphamide dose):

   * ANC ≥1.500 cells/microL o Lymphocyte count ≥ 1.000 cells/microL
   * Platelet count ≥ 100.000 cells/microL
   * Hemoglobin ≥ 9.0 g/dL (patients may be transfused to meet this criterion at least 7 days before).
   * Total bilirubin ≤ 1.5 x ULN (except for patients with known Gilbert's syndrome and serum bilirubin level ≤ 3 x ULN).
   * AST and ALT ≤ 3 x ULN (except for patients with documented liver metastases, in which case AST and ALT is allowed up to ≤ 5 x ULN).
   * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min based on the Cockcroft-Gault glomerular filtration rate estimation.
   * INR ≤ 1.5 x ULN
   * Serum albumin ≥ 25 g/dL
10. Female patient of childbearing potential must have a negative pregnancy test (serum) within 7 days prior to the first study drug administration and agreement to remain abstinent or use of contraceptive measures that result in a failure rate of <1%/year (bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, copper intrauterine devices) during the treatment period or within 12 months after the administration of cyclophosphamide, 7 months after the last dose of trastuzumab, or 6 months after the last dose of pertuzumab, whichever occurs last.

A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a post-menopausal state (>12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of both ovaries and/or uterus).

Patient Exclusion Criteria:

1. Other primary cancers apart from non-melanoma localized skin cancer, carcinoma in situ of the cervix, localized prostate cancer or ductal in situ carcinoma of the breast treated surgically, or prior cancer treated with curative intent at least more than 3 years ago and with no evidence of relapse.
2. Major surgical procedures within 4 weeks prior to the cyclophosphamide dose, or anticipation of need for a major surgical procedure during the course of the study.
3. Less than 3 weeks since last dose of approved systemic anti-cancer therapy (chemotherapy, hormonal therapy, tyrosine kinase inhibitors, immunotherapy, radiotherapy) prior to the cyclophosphamide dose. Less than 6 weeks since last dose of mitomycin C and nitrosoureas. However, non-extended palliative radiotherapy for bone metastases ≤ 2 weeks prior to the cyclophosphamide dose is allowed.
4. Treatment with investigational agent within 4 weeks prior to the cyclophosphamide dose.
5. Prior treatment with adoptive cellular therapy.
6. History of severe allergic, anaphylactic or other hypersensitivity reactions to trastuzumab and/or pertuzumab.
7. Prior G4-3 toxicity to trastuzumab and/or pertuzumab.
8. Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1, except for any grade of alopecia.
9. Administration of a live attenuated vaccine within 4 weeks before the cyclophosphamide dose.
10. Signs or symptoms of systemic infection within 2 weeks prior the cyclophosphamide dose (requiring antibiotics).
11. Patients with active tuberculosis, patients with HIV infection or syphilis, active chronic or acute hepatitis B infection or hepatitis C infection, herpes simplex virus, cytomegalovirus, HTLV or Epstein-Barr virus infection. Patients with prior allogenic bone marrow transplantation or prior solid organ transplantation.
12. Systemic steroid therapy or other immune-suppressants or immune-stimulatory agents (including but not limited to prednisone, azathioprine, methotrexate, thalidomide, anti-TNF agents) within 4 weeks prior to the cyclophosphamide dose.
13. Patients who have received acute, low-dose dexamethasone for nausea, may be enrolled after discussion with the principal investigator.
14. The use of inhaled corticosteroids or mineralocorticoids for orthostatic hypotension/adrenocortical insufficiency (not related with autoimmune disease) is allowed.
15. Corticosteroids as premedication in case of dye allergy prior to imaging tests are allowed.
16. History of autoimmune diseases including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated to antiphospholipid syndrome, granulomatosis, Sjögren's syndrome, multiple sclerosis, vasculitis or glomerulonephritis. Any other potential autoimmune disorders may be accepted after consultation with the principal investigator.

    * Patients with history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
    * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may also be eligible.
17. New York Heart Association (NYHA) functional class ≥ 2, history within the past 6 months of myocardial infarction, unstable angina, coronary artery bypass grafting or stenting, stroke or clinically-significant cardiac arrhythmia (isolated bundle branch blockade in an ECG is not considered relevant).
18. Uncontrolled (persistent) hypertension defined as systolic blood pressure (SBP) >180 mmHg or diastolic blood pressure (DBP) >100 mmHg.
19. LVEF < 50% by echocardiogram or multi-gated acquisition (MUGA) scan.
20. Uncontrolled pleural effusion, pericardial effusion, or ascites that requires recurrent drainage procedures (once monthly or more frequently).
21. Known hereditary or acquired coagulopathies (e.g., hemophilia, von Willebrand's disease, cancer-associated diffuse intravascular coagulation).
22. Concomitant treatment with therapeutic anticoagulants (oral, heparin). Low dose molecular weight heparin for prophylactic purposes is allowed.
23. Current dyspnea at rest due to complications of advanced malignancy or requirement for continuous oxygen therapy.
24. Known primary CNS malignancy or symptomatic or untreated CNS metastases. Patients with asymptomatic or treated CNS metastases may be enrolled after consultation with the Medical Monitor, provided they have improved upon completion of CNS-directed therapy (radiotherapy or surgical removal).
25. Pregnancy or lactation within the past 3 months and throughout the trial.
26. Substance abuse, medical, psychological, or social conditions that may interfere with the subject's participation in the trial or, as per the investigator's judgment, may jeopardize the interpretation of the results or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Nature and frequency of Adverse Events (AE) | From baseline through 6 months from the last dose of IL-2 or until the first dose of the next anticancer therapy, whichever occurs first
Nature and frequency of Serious Adverse Events (SAE) | From baseline through 6 months from the last dose of IL-2 or until the first dose of the next anticancer therapy, whichever occurs first
Treatment-limiting Toxicity (TLT) | From the administration of cyclophosphamide until 28 days after that date.
Alterations in clinical laboratory test results | From baseline through study completion, an average of 24 months
Alterations in ECGs results | From baseline through study completion, an average of 24 months
Alterations in vital sign measurements | From baseline through study completion, an average of 24 months
Alterations in physical examination findings | From baseline through study completion, an average of 24 months
Alterations in assessment of ECOG | From baseline through study completion, an average of 24 months

SECONDARY OUTCOMES:
Overall Response Rate (ORR) (complete response (CR) and partial response (PR)) | From baseline through 6 months from the last dose of IL-2 or until the first dose of the next anticancer therapy, whichever occurs first
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.
Clinical benefit rate (CR + PR + stable disease (SD) at 4-month) assessed by RECIST v.1.1. | From baseline through disease progression, assessed up to 24 months after last dose of IL-2
Duration of response (DOR) by RECIST v1.1. | From baseline through disease progression, assessed up to 24 months after last dose of IL-2
Progression-free survival (PFS). | From baseline through disease progression, assessed up to 24 months after last dose of IL-2
  Defined as the time from the date of first treatment administration to the date of first documentation of disease progression or death due to any cause, whichever occurs first.

OTHER OUTCOMES:
Compare the degree of infiltration of NK, assessed by immunofluorescence (CD56+, CD3-, NKP46+) in the biopsy samples before and after NK infusion. | From baseline to biopsy obtained on Day 3 of treatment
Compare parameters of NK activation: evaluating the activation on apoptotic proteins (e.g. caspase 3) in the biopsy samples before and after NK infusion. | From baseline to biopsy obtained on Day 3 of treatment
Immune cell number and activation will be studied by immunohistochemical methods CD4+ and CD8+ T cells and NK cells) in formalin fixed paraffin embedded (FFPE) tissue. | From baseline to biopsy obtained on Day 3 of treatment
Immune-monitoring of NK numbers and NK phenotype (engraftment of NK from the donor versus patient) in blood, assessed by flow cytometry. | From baseline to Day 21 after trastuzumab/pertuzumab infusion
Chimerism analysis to monitor donor-derived NK cell persistence by PCR | From baseline to biopsy obtained on Day 3 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elena Garralda, MD, Principal Investigator — Vall d'Hebron Institute of Oncology; Ignacio Melero, MD, Principal Investigator — Clinica Universidad de Navarra
Locations (2):
- Spain (2):
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Hospital, Barcelona

IPD SHARING:
Plan to Share IPD: No